CLINICAL TRIAL: NCT03997409
Title: Impact of a Low-Carbohydrate Diet on Glycemic Control and Lipids in Pediatric Type 1 Diabetes
Brief Title: Impact of a Low-Carbohydrate Diet in Pediatric Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sara Duffus, Clinical Fellow, Division of Pediatric Endocrinology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190851
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2022-06

CONDITIONS: Type 1 Diabetes
Keywords: Low Carbohydrate Diet; Standard Carbohydrate Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Carbohydrate Diet (Experimental): The investigators will prescribe isocaloric diets equaling the estimated energy requirements of the Institute of Medicine. Participants on the LCD intervention will consume 25-35% of total daily intake from carbohydrates, 45-65% from fat and 10-30% from protein.
  Interventions: Other: Dietary Intervention
- Standard Carbohydrate Diet (Active Comparator): The investigators will prescribe isocaloric diets equaling the estimated energy requirements of the Institute of Medicine. Participants on the SCD intervention will consume 45-65% of total daily caloric intake from carbohydrates, 25-35% from fat and 10-30% from protein.
  Interventions: Other: Dietary Intervention
- No Dietary Recommendations (No Intervention): This group will serve as a control that receives the same number of education sessions as LCD and SCD group to teach general diabetes management but without specific dietary recommendations.

INTERVENTIONS:
Other: Dietary Intervention — The investigators will prescribe isocaloric diets equaling the estimated energy requirements of the Institute of Medicine with varying macronutrient content in each group.
  Arms: Low Carbohydrate Diet; Standard Carbohydrate Diet

SUMMARY:
Dietary carbohydrate consumption is a key factor influencing postprandial glycemia for patients with type 1 diabetes mellitus (T1DM). Because post-prandial glucose excursions profoundly influence hemoglobin A1c (HbA1c), therapeutic approaches to mitigate post-prandial hyperglycemia are of great importance. The quantity and source of carbohydrates affect post-prandial glycemia more than any other dietary factor. These findings serve as the physiologic basis for a growing interest in carbohydrate-restricted diets in the management of T1DM despite American Diabetes Association (ADA) guidelines that discourage restricting total carbohydrate intake to less than 130 grams per day. Although case series and prospective studies suggest low-carbohydrate diets (LCD) significantly improve HbA1c for adults with T1DM, data in the pediatric T1DM population is limited. The investigators will conduct a randomized prospective pilot study evaluating glycemic control, lipidemia, and quality of life (QOL) in pediatric T1DM patients on a LCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T1DM for at least 12 months
* Age 13 to 21 years
* Total daily dose of insulin 0.5 to 1.25 units/kg/day
* Current use of an insulin pump and CGM
* HbA1c between 7% and 10%
* Tanner stage 3 to 5 on physical exam
* Participant or parent of participant use of smart phone
* Able to read and speak English

Exclusion Criteria:

* Any episode of diabetic ketoacidosis (DKA) in the last 12 months
* Any episode of severe hypoglycemia (defined as requiring assistance from another person, including coma, seizures, or episodes requiring glucagon, IV dextrose or oral carbohydrate administered by another person) in the last 12 months
* Any prior abnormal fasting lipid panel (LDL > 130)
* Additional dietary restrictions
* Following a weight-loss or otherwise restrictive diet
* Use of medication or supplements other than insulin to control blood glucose
* Use of medication or other supplements to lower lipids
* Pregnancy or breast feeding
* History of hemoglobinopathy

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin M Gregory, MD, MSCI, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Started | 14 | 13 | 12
Completed | 10 | 12 | 11
Not Completed | 4 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations | Total
Number analyzed (Participants) | 14 | 13 | 12 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.5 [14.0 to 16.3] | 16 [15.0 to 17.0] | 15.5 [15.0 to 17.0] | 15.5 [14.5 to 16.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 19
  Male | 7 | 7 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 13 | 12 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 13 | 12 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: HbA1c (%) change will be measured from baseline to 12 weeks
Time Frame: Baseline to week 12
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 10 | 12 | 11
percentage | 0.4 [0.1 to 0.4] | 0.3 [-0.2 to 0.5] | -0.2 [-0.3 to 0.2]

2. Secondary Outcome: Percent of Time Spent in the Glycemic Target of 70 - 140 mg/dL
Description: Percent of time is calculated from data collected from the continuous glucose monitor worn by participants. T1DM participants were instructed in the use of a continuous glucose monitor (CGM) for the monitoring of glycemia during the study. Participants were shown how to upload CGM data into a HIPAA and FDA-compliant cloud-based, data-integration platform for analysis.
Time Frame: Baseline to Week 12
Population: Data was not collected for the following participants due to missed study visit: Low Carb Diet: 1 participant; Standard Carb Diet: 1 participant
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
percentage | -3 [-9.2 to 6.2] | -8.9 [-13.0 to 7.2] | 3.4 [0.8 to 10.7]

3. Secondary Outcome: Percent of Time Spent Above the Glycemic Target of 140 mg/dL
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
percentage | -1.4 [-15.8 to 4.5] | -1.9 [-6.1 to 4.4] | -1.9 [-5.3 to 2.7]

4. Secondary Outcome: Percent of Time Spent Below the Glycemic Target of 70 mg/dL
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
percentage | 0 [-0.1 to 1.2] | 0 [-0.3 to 1.2] | -0.2 [-0.4 to 0.3]

5. Secondary Outcome: Percent of Time Spent in Hypoglycemia Below 50 mg/dL
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
percentage | 0 [-0.2 to 0.1] | 0.1 [0 to 0.2] | 0 [-0.2 to 0.2]

6. Secondary Outcome: Change in Average Blood Glucose
Description: Change in average blood glucose is calculated from data collected from the continuous glucose monitor worn by participants. T1DM participants were instructed in the use of a continuous glucose monitor (CGM) for the monitoring of glycemia during the study. Participants were shown how to upload CGM data into a HIPAA and FDA-compliant cloud-based, data-integration platform for analysis.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
mg/dL | 6 [-17 to 14] | 7 [-6 to 25] | -11.5 [-15.5 to -0.5]

7. Secondary Outcome: Change in the Blood Glucose Standard Deviation
Description: Change in the blood glucose standard deviation is calculated from data collected from the continuous glucose monitor worn by participants. T1DM participants were instructed in the use of a continuous glucose monitor (CGM) for the monitoring of glycemia during the study. Participants were shown how to upload CGM data into a HIPAA and FDA-compliant cloud-based, data-integration platform for analysis.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
mg/dL | 0 [-10 to 6] | 0 [-7 to 16] | -3 [-8 to 2]

8. Secondary Outcome: Change in Average Total Daily Dose of Insulin
Description: Average Total Daily Dose of Insulin is calculated from data collected from the the use of an insulin pump by participants. T1DM participants were instructed in the use of an insulin pump for the adminsitration of insulin during the study. Instructions included administering all insulin via insulin pump and recording all carbohydrates consumed into the insulin pump. T1DM participants were instructed how to upload insulin pump data into a HIPAA and FDA-compliant cloud-based, data-integration platform for analysis.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units of insulin/day
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
units of insulin/day | 2.7 [-8.0 to 11.0] | 4.8 [-4.8 to 6.6] | -1.9 [-5.7 to 5.5]

9. Secondary Outcome: Change in Average Bolus Amount of Insulin Per Day
Description: Average bolus amount of Insulin per day is calculated from data collected from the the use of an insulin pump by participants. T1DM participants were instructed in the use of an insulin pump for the adminsitration of insulin during the study. Instructions included administering all insulin via insulin pump and recording all carbohydrates consumed into the insulin pump. T1DM participants were instructed how to upload insulin pump data into a HIPAA and FDA-compliant cloud-based, data-integration platform for analysis.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units of insulin/day
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
units of insulin/day | 3.3 [-7.6 to 11.0] | 5.1 [-6.1 to 7.6] | -1.7 [-5.1 to 2.4]

10. Secondary Outcome: Change in Average Basal Amount of Insulin Per Day
Description: Average Basal Amount of Insulin Per Day is calculated from data collected from the the use of an insulin pump by participants. T1DM participants were instructed in the use of an insulin pump for the adminsitration of insulin during the study. Instructions included administering all insulin via insulin pump and recording all carbohydrates consumed into the insulin pump. T1DM participants were instructed how to upload insulin pump data into a HIPAA and FDA-compliant cloud-based, data-integration platform for analysis.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units of insulin / day
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 9 | 11 | 11
units of insulin / day | 0.2 [-0.1 to 1.8] | -0.2 [-1.6 to 1.3] | 0.2 [-0.8 to 2.9]

11. Secondary Outcome: Change in Low Density Lipoprotein Particle Number
Description: The number of Low Density Lipoprotein Particles (LDL-P) is directly measured using nuclear magnetic resonance (NMR) spectroscopy.
Time Frame: Baseline to 12 weeks
Population: Data was not collected for the following participants due to missed study visit: Low Carb Diet: 2 participants; Standard Carb Diet: 2 participants
Measure: Median (Inter-Quartile Range); unit: Nanomoles per liter (nmol/L)
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 8 | 10 | 11
Nanomoles per liter (nmol/L) | 30 [2.8 to 97.3] | -41 [-76 to 97] | 47 [-25 to 116]

12. Secondary Outcome: Change in High Density Lipoprotein Particle Number
Description: The number of High Density Lipoprotein Particles (HDL-P) is directly measured using nuclear magnetic resonance (NMR) spectroscopy.
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Nanomoles per liter (nmol/L)
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 8 | 10 | 11
Nanomoles per liter (nmol/L) | -1 [-2.2 to 2.4] | 1.5 [-3.2 to 3.0] | -2.3 [-4.2 to 0.3]

13. Secondary Outcome: Change in Small Low Density Lipoprotein Particle Number
Description: The number of Small Low Density Lipoprotein Particles (LDL-P) is directly measured using nuclear magnetic resonance (NMR) spectroscopy.
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Nanomoles per liter (nmol/L)
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 8 | 10 | 11
Nanomoles per liter (nmol/L) | -2.5 [-172.3 to 19.5] | 40 [-49.5 to 78] | -12 [-102 to 31]

14. Secondary Outcome: Change in Low Density Lipoprotein Size
Description: The size of Low Density Lipoprotein Particles (LDL-P) is directly measured using nuclear magnetic resonance (NMR) spectroscopy.
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: nanometer (nm)
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 8 | 10 | 11
nanometer (nm) | 0 [-0.25 to 0.2] | -0.15 [-0.68 to 0.28] | 0.2 [0 to 0.5]

15. Secondary Outcome: Change in Concentration of Serum Ketones (Beta-hydroxybutyrate)
Description: Change is measured by difference in concentration of serum ketones (beta-hydroxybutyrate)
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Millimoles per liter (mmol/L)
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 8 | 10 | 11
Millimoles per liter (mmol/L) | -0.04 [-0.12 to 0.04] | -0.03 [-0.20 to 0.05] | -0.02 [-0.19 to 0.03]

16. Secondary Outcome: Change in Score of Pediatric Quality of Life Inventory (PedsQL) Diabetes Module
Description: The PedsQL 3.0 Teen Report (ages 13-18) is composed of 28 items. Item scaling is a 5-point scale from 0 (never) to 4 (almost always). The total possible range of scores 0-112 Higher scores indicate higher quality of life.
Time Frame: Baseline to week 12
Population: Data was not collected for the following participants due to missed study visit: Low Carb Diet: 3 participants; Standard Carb Diet: 4 participants; No Dietary Recommendations: 2 participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 7 | 8 | 9
units on a scale | -5 [-9 to -1] | -5.5 [-14 to 7.3] | -3 [-7 to -0.5]

17. Secondary Outcome: Change in Diabetes Burden as Measured by the Problem Areas in Diabetes: Teen Version (PAID-T) Report
Description: Diabetes burden was measured using the Problem Areas in Diabetes (PAID-T) parent-report, a measure of how bothersome day-to-day problems are for adolescents with type 1 diabetes. The he PAID-T is a 26 item measure scored on a likert scale from one-to-six with a total possible scale score ranging from 26-156. A lower score represents less burden.
Time Frame: Baseline to week 12
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
Number analyzed (Participants) | 7 | 8 | 9
units on a scale | 3 [-2 to 15] | -5.5 [-11.3 to 10.3] | 4 [-9.5 to 9.5]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | No Dietary Recommendations
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03997409/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03997409/ICF_000.pdf